CLINICAL TRIAL: NCT07137312
Title: MC240903 Ex Vivo Expansion of Tumor Antigen-Specific T Cells for Adoptive T Cell Therapy
Brief Title: Ex Vivo Expansion (ACT-X)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC240903; 24-011832 (Other: Mayo Clinic Institutional Review Board); NCI-2025-06055 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Healthy; Malignant Solid Neoplasm
MeSH Terms: interventions — Blood Specimen Collection; Specimen Handling; Blood Component Removal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained only with participant consent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Blood Draw Group: Participants who elect to provide specimen via standard blood draw. Some participants may provide a specimen via blood draw one time (the "blood draw group") and then elect to provide a second optional specimen via apheresis (the "apheresis group") or vice versa. Thus, which specimen collection group a given participant is in may change based on patient and provider preference for a given visit.
  Interventions: Procedure: Blood Draw; Procedure: Apheresis
- Apheresis Group: Participants who elect to provide specimen via apheresis. Apheresis is a procedure where blood is drawn from the body, specific components like plasma, platelets, and/or white blood cells are separated out, and the rest of the blood is returned. Some participants may provide a specimen via apheresis one time (the "apheresis group") and then elect to provide a second optional specimen via a standard blood draw (the "blood draw group") or vice versa. Thus, which specimen collection group a given participant is in may change based on patient and provider preference for a given visit.
  Interventions: Procedure: Blood Draw; Procedure: Apheresis

INTERVENTIONS:
Procedure: Blood Draw — Participants have a standard blood draw or apheresis on study. Some participants may provide a specimen via apheresis one time (the "blood draw group") and then elect to provide a second optional specimen via a standard blood draw (the "apheresis draw group") or vice versa.
  Other Names: Blood sample collection; Biospecimen collection; Specimen collection
Procedure: Apheresis — Participants have a standard blood draw or apheresis on study. Apheresis is a procedure where blood is drawn from your body, specific components like plasma, platelets, and/or white blood cells are separated out, and the rest of the blood is returned. Some participants may provide a specimen via apheresis one time (the "apheresis group") and then elect to provide a second optional specimen via a standard blood draw (the "blood draw group") or vice versa.

SUMMARY:
The purpose of this study is to understand how the body's immune cells respond to a new type of vaccine (neoantigen vaccine) designed to help the immune system recognize and fight cancer. To do this, the study team will collect a research specimen from participants to study their immune cells' reactions to the neoantigen vaccine. This research will help researchers learn more about how these vaccines might work to protect or treat against cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed current or previous solid malignancy or healthy individuals
* Willing to provide mandatory research blood draw or apheresis per protocol
* Provide written informed consent
* The following laboratory values obtained ≤ 28 days prior to registration

  * Hemoglobin ≥10.0 g/dl
  * Absolute neutrophil count (ANC) ≥1500/mm^3
  * Platelet count ≥100,000/mm^3

Exclusion Criteria:

* Any of the following prior therapies:

  * IV antibiotic ≤2 weeks prior to apheresis
  * Major Surgery ≤4 weeks prior to registration
  * Received a live vaccine ≤30 days prior to registration
* Active hematologic malignancies ≤ 3 years prior to registration
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy
* History of active tuberculosis (TB), human immunodeficiency virus (HIV), active hepatitis B (e.g., HBsAg reactive), and/or active hepatitis C infection [e.g., Hepatitis C Virus (HCV) ribonucleic acid (RNA) qualitative is detected)
* Known history of active autoimmune disease that has required systemic treatment in the ≤14 days (i.e., with the use of disease-modifying agents, corticosteroids >10 mg daily prednisone equivalent, or other immunosuppressive drugs) prior to registration.

  * NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Patients with vitiligo, Graves' disease, or psoriasis not requiring systemic treatment within the past 30 days are not excluded. Patients with Celiac disease controlled with diet modification are not excluded.
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female participants who have/had cancer or are healthy individuals who would like to contribute to cancer research efforts.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Immune effector networks | Baseline; up to 3 years
  Specimen samples obtained by blood draw and/or apheresis will be analyzed to identify immune effector networks that accelerate ex vivo expansion of antigen-specific memory precursor T cells. All tests will be two sided with a p<0.05 being considered as statistically significant.
Dendritic cell signaling programs | Baseline; up to 3 years
  Specimen samples obtained by blood draw and/or apheresis will be analyzed to define dendritic cell signaling programs that foster generation of polyfunctional, high avidity antigen-specific T cells capable of recognizing naturally processed tumor antigen. All tests will be two sided with a p<0.05 being considered as statistically significant.
Cytokine capture methods | Baseline; up to 3 years
  Specimen samples obtained by blood draw and/or apheresis will be analyzed to identify cytokine capture methods for isolation of antigen-specific T cells. All tests will be two sided with a p<0.05 being considered as statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Knutson, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials